CLINICAL TRIAL: NCT01271699
Title: Multiple Sclerosis and Fabry Disease: Prevalence of Fabry Disease in a Defined Population at Risk - Patients Formerly Diagnosed With Multiple Sclerosis - an Epidemiological Study
Brief Title: Prevalence of Fabry Disease in a Defined Population at Risk - Patients Formerly Diagnosed With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: MS01/2011
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2021-04-09 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis
Keywords: Fabry Disease; Fabry´s Disease; Anderson-Fabry Disease; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fabry diagnostic will be done centrally: blood samples will be stored for analysis of a-galactosidase in blood, Gb3 as well as lyso-Gb3. In all cases direct analysis of the gene will be done, especially in females where due to the Lyonisation effect a-galactosidase activity might be normal in blood although the patient might suffer from Fabry disease.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation: Patients at age 18-50 with a confirmed or probably diagnosis of Multiple Sclerosis according to the McDonald diagnostic criteria for MS

SUMMARY:
The association of Multiple Sclerosis (MS) and Fabry disease is known from own clinical experiences as well as from case reports in the literature, where symptoms and suspicious results in the brain MRI led to the misdiagnosis of Fabry patients as MS. Remarkably, those patients almost never showed oligoclonal bands or an intrathecally derived IgG-production was wrongly assumed due to misinterpretation of CSF results. Where oligoclonal bands were present, concomitant diagnoses had to be discussed. Furthermore, those patients showed no involvement of the spinal cord, as evidenced by MRI. Beside the possible complications of a not-effective and not-necessary MS therapy, those patients are at risk of irreparable organ damage due to the delayed implementation of enzyme replacement therapy for Fabry disease.

DETAILED DESCRIPTION:
Fabry disease is an X-linked lysosomal disorder that leads to excessive deposition of neutral glycosphingolipids in the vascular endothelium of several organs in the body. Progressive endothelial accumulation of glycosphingolipids accounts for the associated clinical abnormalities of skin, eye, kidney, heart, brain, and peripheral nervous system. Fabry disease manifesting predominantly in men. Female heterozygotes also present with features of Fabry disease. In Europe the prevalence of Fabry disease seems to be massively underrepresented.

Multiple Sclerosis (MS, Encephalomyelitis disseminata) ist the most common inflammatory disease of the central nervous system (CNS). The first clinical manifestation peaks in the 3rd-4th decade. 2.5 million Young adults are affected worldwide. In Germany the prevalence rate reaches approx. 100 patients per 100,000 inhabitants. Females are more frequently affected (2-3:1). The underlying causes of the disease are not sufficiently explored yet. The genetic backgrounds as well as environmental factors are involved. An autoimmune mediated process, driven by activated T-lymphocytes and macrophages, leads to inflammatory demyelination and axonal loss.

Magnetresonance imaging of the brain and spinal cord, evaluation of the cerebrospinal fluid to detect intrathecally derived immunoglobulin production (IgG) and a comprehensive diagnostic workup on other possible causes of the symptoms. The modern diagnostic criteria (McDonald criteria, 2001 + revisions 2005) demand the proof of the dissemination of the inflammatory process in space and time, either by clinical or radiological terms.

The evaluation of the cerebrospinal fluid aims at the confirmation of an intrathecally derived synthesis of IgG. In 98% of the patients oligoclonal bands can be detected during the course of the disease. This parameter is highly sensitive but only low specific. The diagnostic criteria allow making the diagnosis of "certain" or at least "probable" MS without the confirmation of oligoclonal bands.

ELIGIBILITY:
Inclusion Criteria:

* Patients at age 18-50 years old with a confirmed or probably diagnosis of Multiple Sclerosis according to the McDonald diagnostic criteria for MS
* Patients with confirmed diagnosis of Multiple Sclerosis according to the McDonald diagnostic criteria but without confirmation of oligoclonal IgG in the CSF
* Patients with present oligoclonal IgG in the CSF but without proof of dissemination of spinal inflammatory processes in the MRI
* Signed informed consent

Exclusion Criteria:

* Patients being younger than 18 years or older than 50 years
* Patients without performed MRI of the brain and spinoaxis
* Patients with a structural change in the brain that is not caused by a chronic inflammatory disease of the CNS
* Missing signed informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult Patients at age 18-50 with a confirmed or probably diagnosis of Multiple Sclerosis according to the McDonald diagnostic criteria for Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Fabry Disease in a Defined Population at Risk - Patients Formerly Diagnosed With Multiple Sclerosis | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, MD, Study Chair — CENTOGENE GmbH Rostock

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sims K, Politei J, Banikazemi M, Lee P. Stroke in Fabry disease frequently occurs before diagnosis and in the absence of other clinical events: natural history data from the Fabry Registry. Stroke. 2009 Mar;40(3):788-94. doi: 10.1161/STROKEAHA.108.526293. Epub 2009 Jan 15. PMID 19150871
- [Background] Falke K, Buttner A, Schittkowski M, Stachs O, Kraak R, Zhivov A, Rolfs A, Guthoff R. The microstructure of cornea verticillata in Fabry disease and amiodarone-induced keratopathy: a confocal laser-scanning microscopy study. Graefes Arch Clin Exp Ophthalmol. 2009 Apr;247(4):523-34. doi: 10.1007/s00417-008-0962-9. Epub 2008 Oct 18. PMID 18931853
- [Background] Fellgiebel A, Keller I, Marin D, Muller MJ, Schermuly I, Yakushev I, Albrecht J, Bellhauser H, Kinateder M, Beck M, Stoeter P. Diagnostic utility of different MRI and MR angiography measures in Fabry disease. Neurology. 2009 Jan 6;72(1):63-8. doi: 10.1212/01.wnl.0000338566.54190.8a. PMID 19122032
- [Background] Wang RY, Lelis A, Mirocha J, Wilcox WR. Heterozygous Fabry women are not just carriers, but have a significant burden of disease and impaired quality of life. Genet Med. 2007 Jan;9(1):34-45. doi: 10.1097/gim.0b013e31802d8321. PMID 17224688
- [Background] Rolfs A, Bottcher T, Zschiesche M, Morris P, Winchester B, Bauer P, Walter U, Mix E, Lohr M, Harzer K, Strauss U, Pahnke J, Grossmann A, Benecke R. Prevalence of Fabry disease in patients with cryptogenic stroke: a prospective study. Lancet. 2005 Nov 19;366(9499):1794-6. doi: 10.1016/S0140-6736(05)67635-0. PMID 16298216
- [Background] McDonald WI, Compston A, Edan G, Goodkin D, Hartung HP, Lublin FD, McFarland HF, Paty DW, Polman CH, Reingold SC, Sandberg-Wollheim M, Sibley W, Thompson A, van den Noort S, Weinshenker BY, Wolinsky JS. Recommended diagnostic criteria for multiple sclerosis: guidelines from the International Panel on the diagnosis of multiple sclerosis. Ann Neurol. 2001 Jul;50(1):121-7. doi: 10.1002/ana.1032. PMID 11456302
- [Background] Polman CH, Reingold SC, Edan G, Filippi M, Hartung HP, Kappos L, Lublin FD, Metz LM, McFarland HF, O'Connor PW, Sandberg-Wollheim M, Thompson AJ, Weinshenker BG, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2005 revisions to the "McDonald Criteria". Ann Neurol. 2005 Dec;58(6):840-6. doi: 10.1002/ana.20703. PMID 16283615
- [Background] Rieckmann P, Toyka KV; Multiple Sclerosis Therapy Consensus Group. [Immunomodulatory staged therapy of multiple sclerosis. New aspects and practical applications, March 2002]. Nervenarzt. 2002 Jun;73(6):556-63. doi: 10.1007/s00115-002-1328-x. German. PMID 12243005
- [Background] Callegaro D, Kaimen-Maciel DR. Fabry's disease as a differential diagnosis of MS. Int MS J. 2006 Jan;13(1):27-30. PMID 16420782
- [Background] Saip S, Uluduz D, Erkol G. Fabry disease mimicking multiple sclerosis. Clin Neurol Neurosurg. 2007 May;109(4):361-3. doi: 10.1016/j.clineuro.2006.12.006. Epub 2007 Jan 17. PMID 17234336
- [Background] Invernizzi P, Bonometti MA, Turri E, Benedetti MD, Salviati A. A case of Fabry disease with central nervous system (CNS) demyelinating lesions: a double trouble? Mult Scler. 2008 Aug;14(7):1003-6. doi: 10.1177/1352458508092355. Epub 2008 Jul 16. PMID 18632784